CLINICAL TRIAL: NCT02708823
Title: Standardization of a Novel Self-administered Tablet Computer-based Clinical Screening Tool for Adverse Postoperative Cognitive Outcomes: A Neuropsychological Study in Non-surgical Volunteers
Brief Title: Standardization of a Novel Self-administered Tablet Computer-based Clinical Screening Tool for Adverse Postoperative Cognitive Outcomes
Acronym: CogCheck-Norm
Status: Completed | Type: Observational
Sponsor: Nicolai Goettel (Other)
Responsible Party: Sponsor-Investigator, Nicolai Goettel, MD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: CogCheck-Norm
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Delirium
Keywords: Postoperative delirium; Risk assessment; Clinical screening tool; Tablet computer
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: CogCheck application — The application is administered once to all study participants.

SUMMARY:
Postoperative delirium (POD) and postoperative cognitive dysfunction (POCD) are common complications after surgery and may affect elderly patients in particular. CogCheck, an application for tablet computers, was developed with the intention to assist preoperative risk screening for POD and POCD in surgical patients. The aim of this study is to generate normative data with cognitively healthy participants for the application.

DETAILED DESCRIPTION:
Postoperative delirium (POD) and postoperative cognitive dysfunction (POCD) are common complications after surgery and may affect elderly patients in particular. Prior studies found risk factors for POD and POCD which are present preoperatively, e.g. older age and pre-existing cognitive impairment. However, the preoperative risk of postoperative adverse cognitive outcomes (POD and POCD) is often not screened in routine clinical practice as it is time-consuming and requires trained personnel.

In 2014, the application for tablet computers "Delirium Risk Profile" (DRP) was developed at the University Hospital Basel to assist preoperative screening in surgical patients. The application was later renamed CogCheck as the scope of the tool was extended to POD and POCD risk assessment.

The aim of this study is to provide normative data for the application. Ultimately, the objective is to assist health care providers in the evaluation of patients' cognitive functions by routinely using the application in preoperative clinics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Education ≥ 7 years
* Fluency in the German language
* Written informed consent

Exclusion Criteria:

* History of cognitive impairment
* Signs of depression
* Severe sensory or motor impairment interfering with cognitive testing
* Serious somatic disease, disease or event affecting the central nervous system (head trauma with loss of consciousness > 5 minutes, any brain surgery, general anesthesia within the last 3 months, alcoholism, intoxication with neurotoxic substances)
* Cerebrovascular disease
* Regular medication with psychoactive drugs except for benzodiazepines
* Participation in any cognitive study within the last 3 months or previous participation in a study using the application.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Non-surgical, cognitively healthy volunteers
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
CogCheck | Baseline.
  Score in a self-administered tablet computer-based neuropsychological assessment.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Baseline.
  Obtained score in MMSE.
Geriatric Depression Scale (GDS) | Baseline.
  Obtained score in GDS.
Consortium to Establish a Registry for Alzheimer's Disease - Neuropsychological Assessment Battery (CERAD-NAB) | Baseline.
  Obtained score in CERAD-NAB.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Goettel, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
No.